CLINICAL TRIAL: NCT01160393
Title: Atrial Fibrillation After Cardiac Surgery - Prospective, Randomized Study Comparing Conventional and Miniaturized Bypass Systems
Brief Title: Atrial Fibrillation After Cardiac Surgery-comparing Conventional and Miniaturized Bypass Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KUH5070216
Record Dates: First submitted 2010-07-05; First posted 2010-07-12 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Cardiac surgery; Prevention; Conventional bypass system; Miniaturized bypass system; Arrhythmia; The Incidence of atrial fibrillation after cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Miniaturized bypass system (Other): Miniaturized bypass system and the incidence of atrial fibrillation after cardiac surgery
  Interventions: Device: Miniaturized bypass system

INTERVENTIONS:
Device: Miniaturized bypass system — Compare the conventional bypass system and miniaturized bypass system of the incidence of atrial fibrillation after cardiac surgery
  Other Names: Miniaturized extracorporeal circulation

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia after cardiac surgery. The incidence of AF varies between 20 - 45 % after (coronary artery bypass grafting) CABG. It may lead to hemodynamic compromise, thromboembolic events, increased length of stay in the hospital and increased morbidity. The underlying cause of AF has been related to a variety of factors. Those most commonly related to the intraoperative management are the use of cardiopulmonary bypass (CPB), the influence of systemic inflammation, myocardial damage, intraoperative fluid management and the need of red blood cell transfusion.

The purpose of the study is to find out the difference in the incidence of atrial fibrillation after CABG when using the conventional (CECC) or mini bypass system (MECC).

The treatment protocol is similar in both groups except the CPB method (CECC vs. MECC). In both methods the investigators use MAQUET tubing and oxygenator. The investigators also collect special blood samples for determining most relevant factors found affecting in the incidence of AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia after cardiac surgery. The incidence of AF varies between 20 - 45 % after (coronary artery bypass grafting) CABG. It may lead to hemodynamic compromise, thromboembolic events, increased length of stay in the hospital and increased morbidity. The underlying cause of AF has been related to a variety of factors. Those most commonly related to the intraoperative management are the use of cardiopulmonary bypass (CPB), the influence of systemic inflammation, myocardial damage, intraoperative fluid management and the need of red blood cell transfusion.

The purpose of the study is to find out the difference in the incidence of atrial fibrillation after CABG when using the conventional (CECC) or mini bypass system (MECC). There has been some evidence in retrospective studies comparing conventional and mini bypass systems that the incidence of AF after mini bypass could be statistically lower.

With the prospective randomized study protocol patient demographic will be similar regarding other variables such as age, gender, previous history of AF, use of beta blockers etc. Only isolated CABG procedures will be included. The amount of patients needed in the study has been calculated so that when the investigators assume that the incidence of AF is normally 45 % and with the mini bypass system the investigators can reduce it to 25 %, the investigators need 330 patients (165 in each group) to show this with the power of 0,8 (a 0,05).

The treatment protocol is similar in both groups except the CPB method (CECC vs. MECC). In both methods the investigators use MAQUET tubing and oxygenator. Fluid management and the use of inotropic agents are standardized and followed by using pulmonary artery catheter. After the operation in the ICU the investigators also use a standardized treatment protocol in the fluid management and in the medication. Patients are ECG-monitored 48 hours after the operation. Possible arrhythmias are documented until the patient is discharged from the hospital.

The investigators also collect special blood samples for determining most relevant factors found affecting in the incidence of AF (IL-6, IL-8, PAI-1).

ELIGIBILITY:
Inclusion Criteria:

* Elective CABC patients

Exclusion Criteria:

* Previous episodes of AF of flutter
* Contraindications for betablocker use
* Sick sinus syndrome
* II or III degree atrioventricular block
* Uncontrolled heart failure
* Previous medication of corticosteroids and immunosuppressive medication
* Emergency surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation | up to 10 days
  The primary endpoint of this study is the incidence of atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Korvenoja, MD, Principal Investigator — Cardiac anesthesiologist, KuopioUH
Locations (1):
- Kuopio University Hospital, Kuopio, Finland